CLINICAL TRIAL: NCT02080442
Title: Balance Training for COPD in Pulmonary Rehabilitation (PR): An Effectiveness Study
Brief Title: Balance Training for Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: Samantha Harrison (Other)
Collaborators: Ontario Lung Association (Other)
Responsible Party: Sponsor-Investigator, Samantha Harrison, Ms Samantha Harrison, West Park Healthcare Centre
Organization: West Park Healthcare Centre (Other)
Other Study IDs: 13-o11-WP
Record Dates: First submitted 2014-03-03; First posted 2014-03-06 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Balance; Pulmonary Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Chronic Obstructive Pulmonary Disease
  Interventions: Other: Balance training

INTERVENTIONS:
Other: Balance training — Training will consist of 30 minute sessions 2-3 times/week for a total of 18-24 sessions, in keeping with best practice guidelines for older adults.12 Sessions will be supervised by physical therapists, using a circuit training approach with different stations designed to target specific areas of impairment. Participants will work through stations in a group setting; however, will receive individualized exercise prescription regarding level of difficulty and exercise progression.

SUMMARY:
The study will involve direct knowledge translation of a laboratory-based study of balance training for patients with COPD, first to the investigators PR program and then, after disseminating the results, this approach could be used to impact on clinical practice in any PR program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* Self-report of decline in balance or fall in the last 5 years or a recent near fall
* Smoking history greater than 10 pack years
* Are able to provide written informed consent.

Exclusion Criteria:

* An inability to communicate because of language skills, hearing or cognitive impairment
* Evidence of a neurological or musculoskeletal condition that severely limits mobility and postural control (e.g., cerebrovascular accident, advanced Parkinson's disease, amputation).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with COPD enrolled in PR
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2013-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | at 6 weeks
  The BBS was assessed following completion of the balance training which took place thrice weekly for a period of 6 weeks.
Timed Up and Go (TUG): | at 6 weeks
  The TUG was assessed following completion of the balance training which took place thrice weekly for a period of 6 weeks.

SECONDARY OUTCOMES:
The Balance Evaluation Systems Test (BESTest) | at 6 weeks
  The BESTest was assessed following completion of the balance training which took place thrice weekly for a period of 6 weeks.
Activity-specific Balance Confidence (ABC) Scale | at 6 weeks
  The ABC scale was assessed following completion of the balance training which took place thrice weekly for a period of 6 weeks.

OTHER OUTCOMES:
Balance training progression: the training prescription and progression will be recorded | at 6 weeks
Therapists' and the participants' satisfaction | at 6 weeks
  Patients completed a questionnaire following completion of the balance training which took place thrice weekly for a period of 6 weeks.
  The focus group was conducted at the end of study recruitment.
Safety: any adverse events associated with balance training will be recorded | at 6 weeks
Applicability and adherence | at 6 weeks
The Six-Minute Walk Test (6MWT) | at 6 weeks
  The 6MWT was assessed by the physiotherapists responsible for delivering the PR program. The PR programs runs over 6 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- West Park Healthcare Center, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Harrison SL, Beauchamp MK, Sibley K, Araujo T, Romano J, Goldstein RS, Brooks D. Minimizing the evidence-practice gap - a prospective cohort study incorporating balance training into pulmonary rehabilitation for individuals with chronic obstructive pulmonary disease. BMC Pulm Med. 2015 Jul 23;15:73. doi: 10.1186/s12890-015-0067-2. PMID 26202647